CLINICAL TRIAL: NCT04110288
Title: Vascular Quality Initiative (VQI) - Data Extraction and Longitudinal Trend Analysis (DELTA) Paclitaxel Device Safety Analysis - Phase I Study
Brief Title: VQI DELTA Paclitaxel Device Safety Analysis
Acronym: VQI-PTX
Status: Completed | Type: Observational
Sponsor: Lahey Clinic (Other)
Collaborators: Society for Vascular Surgery Patient Safety Organization (Other)
Responsible Party: Principal Investigator, Frederic S. Resnic, Chair - Division of Cardiovascular Medicine, Lahey Clinic
Other Study IDs: 20193123; U01FD004963 (FDA)
Record Dates: First submitted 2019-09-27; First posted 2019-10-01 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Peripheral Vascular Disease
MeSH Terms: conditions — Peripheral Vascular Diseases | interventions — Paclitaxel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Uncoated Balloon Treatment: Patients treated for PAD with balloon angioplasty, without use of stent.
  Interventions: Device: Non-drug coated Device Treatment
- Bare Metal Stent Treatment: Patients treated for PAD with implantation of bare metal stent.
  Interventions: Device: Non-drug coated Device Treatment
- Paclitaxel Coated Balloon: Patients treated for PAD with drug coated balloon angioplasty, without use of stent.
  Interventions: Drug: Paclitaxel
- Paclitaxel Eluting Stent: Patients treated for PAD with implantation of Paclitaxel DES.
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel to treat peripheral arterial disease
  Other Names: Taxol
  Groups: Paclitaxel Coated Balloon; Paclitaxel Eluting Stent
Device: Non-drug coated Device Treatment
  Groups: Bare Metal Stent Treatment; Uncoated Balloon Treatment

SUMMARY:
The VQI-DELTA Paclitaxel Device Safety Analysis seeks to assess the comparative safety of paclitaxel coated balloons and stents in the treatment of peripheral artery disease (PAD) through analysis of the VQI Peripheral Vascular Intervention (PVI) registry module using the DELTA system.

DETAILED DESCRIPTION:
The VQI-DELTA Paclitaxel Device Safety Analysis seeks to assess the comparative safety of paclitaxel coated balloons and stents in the treatment of PAD through analysis of the Vascular Quality Initiative (VQI) Peripheral Vascular Intervention (PVI) registry module using the DELTA system.

The objective of the VQI - DELTA Paclitaxel Phase I Study is to evaluate the relative safety of Paclitaxel used as an antiproliferative agent in the treatment of symptomatic PAD. The study will analyze Paclitaxel Drug Coated Balloons (DCB) and Paclitaxel Drug Eluting Stents (DES), both together and as unique exposures using propensity score matched survival analysis. If a mortality signal is detected, factors associated with late mortality will be further explored. Phase I is the retrospective component of the planned study, evaluating the 2-year survival of patients treated with a paclitaxel containing/eluting device to matched patients treated with non-paclitaxel devices for symptomatic PAD.

All proposed analyses will be performed using DELTA v3.x, which has the capability to prospectively monitor clinical data repositories for safety signals, and is designed to support risk-adjusted prospective safety surveillance analyses of complex clinical datasets.

Three principle analyses are planned:

1. Paclitaxel DCB (including the Bard Lutonix, Medtronic In.Pact and Philips Spectranetics Stellarex DCB's) as compared with propensity matched patients treated with plain balloons.
2. Paclitaxel delivering DES (including the Cook Zilver PTX and Boston Scientific Eluvia DES) as compared with propensity matched cases using bare metal stents (BMS).
3. Patients treated with either Paclitaxel DCB or Paclitaxel DES compared with propensity matched controls (with DCB patients matched to patients treated with plain balloons, and DES patients matched to patients treated with BMS).

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent endovascular interventional treatment of the femoral or popliteal arteries for symptomatic Peripheral Artery Disease.

Exclusion Criteria:

* In an effort to focus this safety evaluation on those patients being treated in accordance with accepted 'best practice' endovascular intervention strategies and 'on-label' use of devices, patients will be excluded from either exposure cases or controls if they received a balloon expandable stent or a balloon expandable stent graft in the treatment of femoral or popliteal disease. Balloon expandable stents were excluded because these stents have historically shown inferior patency and current best practice favors placement of self-expanding nitinol stents which were engineered for the femoral popliteal segment and tested in multiple trials for this indication 12-14.

Additionally, patients will be excluded (as either potential cases or controls) if their index procedure was performed for acute limb ischemia due to the different etiologies (embolism, in-situ thrombosis) as compared with chronic conditions as they have different treatment paradigms and higher major amputation and mortality rates.

In addition, patients with prior angioplasty or stenting of the superficial femoral artery (SFA)-popliteal segment will be excluded in order to avoid the possibility of improperly assigning paclitaxel exposure to the control group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients, age 18 or older, who underwent endovascular interventional treatment of the femoral or popliteal arteries for symptomatic PAD between 1/1/17 through 4/1/2020 will be candidates for inclusion in the analyses.
Sampling Method: Probability Sample
Enrollment: 219483 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Survival from Death | 2 years post intervention
  Freedom from death of any cause

SECONDARY OUTCOMES:
Intervention Success | 2 year post intervention
  Freedom from death (any cause), re-treatment or major amputation
Successful Ambulation | 1 year post intervention
  Successfully ambulating, ambulating with assistance or with prosthesis

OTHER OUTCOMES:
Falsification - Freedom from Resuming Smoking | 2 year post intervention
  Not resuming smoking post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Frederic S Resnic, MD MSc, Principal Investigator — Lahey Hospital & Medical Center; Daniel Bertges, MD, Study Chair — Society for Vascuar Surgery Patient Safety Organization; Jens Eldrup-Jorgensen, MD, Study Director — Society for Vascuar Surgery Patient Safety Organization
Locations (1):
- Lahey Clinic, Inc., Burlington, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Katsanos K, Spiliopoulos S, Kitrou P, Krokidis M, Karnabatidis D. Risk of Death Following Application of Paclitaxel-Coated Balloons and Stents in the Femoropopliteal Artery of the Leg: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Am Heart Assoc. 2018 Dec 18;7(24):e011245. doi: 10.1161/JAHA.118.011245. PMID 30561254
- [Background] Resnic FS, Majithia A, Marinac-Dabic D, Robbins S, Ssemaganda H, Hewitt K, Ponirakis A, Loyo-Berrios N, Moussa I, Drozda J, Normand SL, Matheny ME. Registry-Based Prospective, Active Surveillance of Medical-Device Safety. N Engl J Med. 2017 Feb 9;376(6):526-535. doi: 10.1056/NEJMoa1516333. Epub 2017 Jan 25. PMID 28121489
- [Background] Kumar A, Matheny ME, Ho KK, Yeh RW, Piemonte TC, Waldman H, Shah PB, Cope R, Normand SL, Donnelly S, Robbins S, Resnic FS. The data extraction and longitudinal trend analysis network study of distributed automated postmarket cardiovascular device safety surveillance. Circ Cardiovasc Qual Outcomes. 2015 Jan;8(1):38-46. doi: 10.1161/CIRCOUTCOMES.114.001123. Epub 2014 Dec 9. PMID 25491915
- [Background] Resnic FS, Gross TP, Marinac-Dabic D, Loyo-Berrios N, Donnelly S, Normand SL, Matheny ME. Automated surveillance to detect postprocedure safety signals of approved cardiovascular devices. JAMA. 2010 Nov 10;304(18):2019-27. doi: 10.1001/jama.2010.1633. PMID 21063011
- [Background] Schillinger M, Minar E. Past, present and future of femoropopliteal stenting. J Endovasc Ther. 2009 Feb;16 Suppl 1:I147-52. doi: 10.1583/1545-1550-16.16.I-147. PMID 19317587
- [Background] Dick P, Wallner H, Sabeti S, Loewe C, Mlekusch W, Lammer J, Koppensteiner R, Minar E, Schillinger M. Balloon angioplasty versus stenting with nitinol stents in intermediate length superficial femoral artery lesions. Catheter Cardiovasc Interv. 2009 Dec 1;74(7):1090-5. doi: 10.1002/ccd.22128. PMID 19859954
- [Background] Chowdhury MM, McLain AD, Twine CP. Angioplasty versus bare metal stenting for superficial femoral artery lesions. Cochrane Database Syst Rev. 2014 Jun 24;2014(6):CD006767. doi: 10.1002/14651858.CD006767.pub3. PMID 24959692
- [Background] Eliason JL, Wainess RM, Proctor MC, Dimick JB, Cowan JA Jr, Upchurch GR Jr, Stanley JC, Henke PK. A national and single institutional experience in the contemporary treatment of acute lower extremity ischemia. Ann Surg. 2003 Sep;238(3):382-9; discussion 389-90. doi: 10.1097/01.sla.0000086663.49670.d1. PMID 14501504
- [Background] Earnshaw JJ, Whitman B, Foy C. National Audit of Thrombolysis for Acute Leg Ischemia (NATALI): clinical factors associated with early outcome. J Vasc Surg. 2004 May;39(5):1018-25. doi: 10.1016/j.jvs.2004.01.019. PMID 15111854
- [Background] Howard DP, Banerjee A, Fairhead JF, Hands L, Silver LE, Rothwell PM; Oxford Vascular Study. Population-Based Study of Incidence, Risk Factors, Outcome, and Prognosis of Ischemic Peripheral Arterial Events: Implications for Prevention. Circulation. 2015 Nov 10;132(19):1805-15. doi: 10.1161/CIRCULATIONAHA.115.016424. Epub 2015 Sep 8. PMID 26350058
- [Background] Baril DT, Ghosh K, Rosen AB. Trends in the incidence, treatment, and outcomes of acute lower extremity ischemia in the United States Medicare population. J Vasc Surg. 2014 Sep;60(3):669-77.e2. doi: 10.1016/j.jvs.2014.03.244. Epub 2014 Apr 24. PMID 24768362
- [Background] Gerhard-Herman MD, Gornik HL, Barrett C, Barshes NR, Corriere MA, Drachman DE, Fleisher LA, Fowkes FGR, Hamburg NM, Kinlay S, Lookstein R, Misra S, Mureebe L, Olin JW, Patel RAG, Regensteiner JG, Schanzer A, Shishehbor MH, Stewart KJ, Treat-Jacobson D, Walsh ME. 2016 AHA/ACC Guideline on the Management of Patients With Lower Extremity Peripheral Artery Disease: Executive Summary: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. J Am Coll Cardiol. 2017 Mar 21;69(11):1465-1508. doi: 10.1016/j.jacc.2016.11.008. Epub 2016 Nov 13. No abstract available. PMID 27851991
- [Background] Hsieh FY, Lavori PW, Cohen HJ, Feussner JR. An overview of variance inflation factors for sample-size calculation. Eval Health Prof. 2003 Sep;26(3):239-57. doi: 10.1177/0163278703255230. PMID 12971199
- [Background] Cepeda MS, Boston R, Farrar JT, Strom BL. Comparison of logistic regression versus propensity score when the number of events is low and there are multiple confounders. Am J Epidemiol. 2003 Aug 1;158(3):280-7. doi: 10.1093/aje/kwg115. PMID 12882951
- [Background] Vidi VD, Matheny ME, Resnic FS. Post-marketing device safety surveillance. Contemp Clin Trials. 2011 May;32(3):307-8. doi: 10.1016/j.cct.2011.02.002. Epub 2011 Feb 28. No abstract available. PMID 21371573
- [Background] Austin PC. Optimal caliper widths for propensity-score matching when estimating differences in means and differences in proportions in observational studies. Pharm Stat. 2011 Mar-Apr;10(2):150-61. doi: 10.1002/pst.433. PMID 20925139
- [Background] Oakes D, Feng C. Combining stratified and unstratified log-rank tests in paired survival data. Stat Med. 2010 Jul 20;29(16):1735-45. doi: 10.1002/sim.3921. PMID 20572124
- [Derived] Bertges DJ, Eldrup-Jorgensen J, Robbins S, Ssemaganda H, Malone M, Marinac-Dabic D, Smale J, Lottes AE, Majithia A, Resnic FS; Society for Vascular Surgery Vascular Quality Initiative. Vascular Quality Initiative Surveillance of Femoropopliteal Artery Paclitaxel Devices. JACC Cardiovasc Interv. 2021 Dec 13;14(23):2598-2609. doi: 10.1016/j.jcin.2021.08.058. PMID 34887051

DOCUMENTS (1):
  • Study Protocol (2020-05-20): https://cdn.clinicaltrials.gov/large-docs/88/NCT04110288/Prot_001.pdf